CLINICAL TRIAL: NCT03798912
Title: A Phase 1 Study of the Safety and Pharmacokinetics of Single Doses of Octreotide Administered Orally Via the RaniPill™ Capsule in Healthy Subjects
Brief Title: A First-in-Human Study of the RaniPill, an Oral Drug Delivery Platform
Acronym: RaniPill
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RANI Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TST-0114
Record Dates: First submitted 2018-12-13; First posted 2019-01-10 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Healthy Volunteers
Keywords: RaniPill capsule, drug delivery, octreotide, pharmacokinetic

STUDY DESIGN:
Intervention Model Description: Healthy men and women volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (4):
- Intravenous octreotide group (Active Comparator): Octreotide 100 mcg will be injected intravenously and serial blood samples will be collected for PK analysis
  Interventions: Combination Product: RaniPill capsule containing octreotide
- RaniPill A group (Experimental): In 20 subjects, a RaniPill with a small balloon size will be administered and serial blood samples will be collected for PK analysis
  Interventions: Combination Product: RaniPill capsule containing octreotide
- RaniPill B group (Experimental): In 20 subjects, a RaniPill with a larger balloon size will be administered and serial blood samples will be collected for PK analysis
  Interventions: Combination Product: RaniPill capsule containing octreotide
- RaniPill C group (Experimental): In 20 subjects, a RaniPill with a different size will be administered and blood samples will be collected for the presence of drug
  Interventions: Combination Product: RaniPill capsule containing octreotide

INTERVENTIONS:
Combination Product: RaniPill capsule containing octreotide — Administration of a RaniPill capsule loaded with 100 mcg of octreotide. Serial blood samples will be collected over the following 4 h for pharmacokinetic analysis of octreotide a) injected intravenously and b) delivered directly into the jejunal wall by the RaniPill capsule.

SUMMARY:
The objective of this study is to ascertain the safety, tolerability and performance of the RaniPill capsule in healthy volunteers

DETAILED DESCRIPTION:
The RaniPill device is capsule-like ingestible device, which injects a microneedle containing a microtablet (payload/drug) into the intestinal wall. This is a phase I (first-in-human) open-label study in healthy volunteers. In 6 subjects, 100 mcg of octreotide (Sandostatin®) will be injected intravenously. Three versions of the RaniPill (A, B and C) will be tested in additional three groups of healthy volunteers (N=20 each). All devices will contain 100 mcg of octreotide. The bioavailability of octreotide will be determined by serial blood sampling in Groups A and B. Performance of the RaniPill will be evaluated in all groups.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form
* Willing to comply with all study procedures and available for the entire duration of the study
* Age between 18 and 55 years
* BMI 17 - 32 kg/m2
* In good general health confirmed by medical history, physical examination, and absence of clinically important laboratory abnormalities per investigator's judgment;
* Women of reproductive potential must use, between study day and the final study visit, a highly effective contraceptive, as defined in the Informed Consent Document, and have a negative urine pregnancy test at the time of screening, as well as on the day of study.

Exclusion Criteria:

* Unable to swallow an intact 000 capsule with water
* History of gastrointestinal surgery or illness, including diarrhea, constipation or other manifestations suggestive of abnormal digestion
* Use of an antacid, proton pump inhibitor or histamine H2 receptor antagonist within 5 days of study day
* Barium ingestion within 30 days of study day
* Allergy or sensitivity to contrast media, iodine, barium sulfate, or latex
* History chronic disease other than mild to moderate systemic hypertension
* Menstruation on day of dosing
* Pregnancy or lactating state
* Participation in an investigational or marketed drug trial within 30 days of the screening visit
* Low likelihood, in the investigator's judgment, to complete the study as required per study plan;
* Any other history which, in the investigator's judgment, makes the subject ineligible or exposes the subject to a risk;
* History of allergic reactions to a component of the RaniPill device or any allergic history other than common food (i.e. shellfish) or insect (i.e. bees) allergies;
* Febrile illness within 5 days;
* History of drug or alcohol abuse or any other factor that, in the investigator's opinion, may interfere with the subject's ability to cooperate and comply with the study procedures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

PRIMARY OUTCOMES:
Incidence and kind of adverse events possibly related to the RaniPill capsule | Up to 30 days after ingestion of the device
  All adverse events possibly related to the device, including abdominal pain, nausea and vomiting, injuries to the gastrointestinal tract and abnormal changes in blood tests results will be monitored and recorded

SECONDARY OUTCOMES:
Pharmacokinetic profile of octreotide delivered by the RaniPill capsule | 4 to 8 hours
  Measurements of octreotide concentration in plasma samples collected serially over 4 h following the deployment of the RaniPill
Confirmation of the excretion of all RaniPill device components | up to 7 days
  Stool examinations to verify that all components of the RaniPill capsule have been defecated

CONTACTS AND LOCATIONS:
Overall Officials: Arvinder K Dhalla, PhD, Study Director — RANI Therapeutics
Locations (1):
- Nucleus Network, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No